CLINICAL TRIAL: NCT03390452
Title: Mobile Phone Messaging to Parents: To Improve Oral Hygiene Among Primary School Children In Quetta, Pakistan
Brief Title: Mobile Phone Messaging To Improve Oral Hygiene Among Primary School Children in Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Services Academy, Islamabad, Pakistan (Other)
Responsible Party: Principal Investigator, Dr. Ashfaq Ahmed Khawaja Khail, PhD Fellow (Public Health), Health Services Academy, Islamabad, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2212-HSA/Ph.D-2015
Record Dates: First submitted 2016-08-11; First posted 2018-01-04 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Oral Hygiene; Dental Plaque Induced Gingivitis
Keywords: mHealth; Oral Health; Primary School Children; Mobile Phone Messaging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The parents will receive "Mobile phone messages" about oral hygiene and healthy dieting of their children through teachers.
  The message format will be text and images, depending upon the education/ literacy level of the parents. Parents will be reminded and information reinforced, at frequent intervals for a period of six months.
  Oral hygiene of School children will be assessed before intervention, after 6 months interval
  Interventions: Behavioral: Mobile Phone Messaging
- Control (No Intervention): The primary school children in the control group will not receive any intervention via their parents or teachers (in-active controls) but will be observed on selected outcome measures for baseline data, then at six month interval to compare for differences (if any) with intervention group.

INTERVENTIONS:
Behavioral: Mobile Phone Messaging — Parents of primary school children will receive "Mobile Phone Messages" regarding their children's oral hygiene maintenance and their positive dietary habits.
  Arms: Intervention

SUMMARY:
Oral health is an important component of general health and oral cavity acts as a mirror to the health of individuals and communities. Inadequate focus on primary prevention of oral diseases, poses a sizeable challenge for numerous countries, especially low and middle income countries.

Mobile phone technology is relatively new and its successes in chronic disease is well documented but there is little evidence available in its use for improving oral health and dietary habits of children.

This will be a Pilot Randomized Control Trial (RCT) . It will be conducted in public and private sector schools of Quetta city, Pakistan. Study will comprise of intervention and a control arm. Duration of intervention is 6 months.

In the intervention group, study participants will be the parents. School teachers will send oral health education and reminder messages on frequent intervals to educate children's parents on oral hygiene and reinforce their behaviors to improve their child oral health.

The primary school children in the control group will not receive any intervention

DETAILED DESCRIPTION:
Oral health is a vital part of general health and oral cavity is considered as a mirror to the health of individuals and communities. Poor oral health has a great impact on general health and several oral conditions are found to be associated with heart and lung diseases, diabetes, low-birth-weight and premature births. Oral conditions also affect the quality of life through affecting speech, eating, education, facial appearance, confidence and social interaction.

Schools settings are important to reach children. School going age is considered as a receptive and influential phase in an individual's life during which lifelong health related behaviors, attitudes and beliefs are developed. Parents have great role in improving their children's oral health. They can influence their children oral health and behaviors and can provide a supportive environment to their children at home in terms of oral hygiene and diet and prevention of risk factors for oral diseases.

Mobile phone text messaging is a powerful tool for changing behaviors as these are common, available, low-cost, and quick.(30) Text messaging can be utilized in reducing the global burden of diseases by promoting healthy behaviors and supporting disease prevention

The main objective of this study is to assess the use of mobile phone (health) messages to Parents of public and private sector primary school children to improve their oral hygiene status

This study will be a Pilot Randomized Control Trial (RCT), comprising of two arms Intervention and Control arm.

In the intervention groups study participants will be the school teachers, parents and primary school children. School teachers will be provided messages (designed by Dental Public Health Professionals or adopted from other sources) through the researcher himself. The teachers will then form groups to send oral health education and reminder messages on frequent intervals to educate children's parents on oral hygiene and reinforce their behaviors to improve their child oral health. Parents will receive mobile phone messages about oral hygiene and healthy dieting of their children by the teachers. The message format will be text and images, depending upon the education/ literacy level of the parents. Parents will be reminded and information reinforced, at frequent intervals for a period of six months. School Children will be evaluated on their oral hygiene through gingival bleeding and plaque scores at the start of intervention, after three months and at the end of intervention i.e six months.

The primary school children in the control group will not receive any intervention via their parents or teachers (in-active controls) but will be observed on selected outcome measures for baseline data, then at 3 months and at six month interval to compare for differences (if any) with intervention group.

The total duration of this study is two years (2017 to 2018) including the intervention which will be of six months duration.

After six months of start of intervention; both the intervention group and the control group will be assessed and evaluated on the primary outcome i.e. Oral hygiene measured through "Oral Hygiene Index" which is a standardized index for assessing oral hygiene and recommended by World health Organization.

ELIGIBILITY:
Inclusion Criteria:

* School children enrolled in primary schools (public and private) in Quetta city.
* Primary School children who are permanent residents of Quetta

Exclusion Criteria:

* Primary School children whose parents/caregivers do not own a mobile phone
* Primary School children having orthodontic or any other mouth appliance for example Braces etc.
* Primary School children who have been diagnosed for a systemic illness e.g. Blood disorders or, Diabetes
* Primary School children who are absent during the time of data collection

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 362 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change in the Oral Hygiene Index Scores | 6 months
  Oral hygiene will be measured through "Simplified Oral Hygiene Index" (OHI-S). Each participant will undergo a dental examination in the school by a trained group of examiners (Qualified Dentists). The WHO recommended protocols for Dental examinations will be followed in assessing outcome measure.
  Simplified Oral Hygiene Index (OHI-S) was developed by Greene and Vermillion in 1964. The OHI-S has two components, the Debris Index (DI) and the Calculus Index (CI). Each of these indexes is based on numerical determinations representing the amount of debris or calculus found on the pre-selected tooth surfaces. For each individual, the debris scores are totaled and divided by the number of surfaces scored. The average individual or group debris and calculus scores are combined to obtain the "Simplified Oral Hygiene Index".
  The group baseline scores for both the arms will be compared with the post-intervention scores to observe the change (if any) to conclude the study results

CONTACTS AND LOCATIONS:
Overall Officials: Ashfaq A Khawajakhail, MPH, Principal Investigator — Health services Academy, Islamabad
Locations (2):
- Pakistan (2):
  - Ashfaq Ahmed Khawajakhail, Quetta, Balochistan
  - Dental Section, Sandman Provincial Hospital Quetta, Quetta, Balochistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Petersen PE. The World Oral Health Report 2003: continuous improvement of oral health in the 21st century--the approach of the WHO Global Oral Health Programme. Community Dent Oral Epidemiol. 2003 Dec;31 Suppl 1:3-23. doi: 10.1046/j..2003.com122.x. PMID 15015736
- [Background] Higgs ES, Goldberg AB, Labrique AB, Cook SH, Schmid C, Cole CF, Obregon RA. Understanding the role of mHealth and other media interventions for behavior change to enhance child survival and development in low- and middle-income countries: an evidence review. J Health Commun. 2014;19 Suppl 1(sup1):164-89. doi: 10.1080/10810730.2014.929763. PMID 25207452
- [Background] Kay E, Locker D. A systematic review of the effectiveness of health promotion aimed at improving oral health. Community Dent Health. 1998 Sep;15(3):132-44. PMID 10645682
- [Background] Ben-Zeev D, Schueller SM, Begale M, Duffecy J, Kane JM, Mohr DC. Strategies for mHealth research: lessons from 3 mobile intervention studies. Adm Policy Ment Health. 2015 Mar;42(2):157-67. doi: 10.1007/s10488-014-0556-2. PMID 24824311
- [Background] Watt RG. Strategies and approaches in oral disease prevention and health promotion. Bull World Health Organ. 2005 Sep;83(9):711-8. Epub 2005 Sep 30. PMID 16211164
- [Background] Haleem A, Siddiqui MI, Khan AA. School-based strategies for oral health education of adolescents--a cluster randomized controlled trial. BMC Oral Health. 2012 Dec 18;12:54. doi: 10.1186/1472-6831-12-54. PMID 23249443
- [Background] Saied-Moallemi Z, Virtanen JI, Vehkalahti MM, Tehranchi A, Murtomaa H. School-based intervention to promote preadolescents' gingival health: a community trial. Community Dent Oral Epidemiol. 2009 Dec;37(6):518-26. doi: 10.1111/j.1600-0528.2009.00491.x. Epub 2009 Aug 20. PMID 19694774
- [Background] da Costa TM, Barbosa BJ, Gomes e Costa DA, Sigulem D, de Fatima Marin H, Filho AC, Pisa IT. Results of a randomized controlled trial to assess the effects of a mobile SMS-based intervention on treatment adherence in HIV/AIDS-infected Brazilian women and impressions and satisfaction with respect to incoming messages. Int J Med Inform. 2012 Apr;81(4):257-69. doi: 10.1016/j.ijmedinf.2011.10.002. Epub 2012 Jan 31. PMID 22296762
- [Background] Park LG, Howie-Esquivel J, Dracup K. A quantitative systematic review of the efficacy of mobile phone interventions to improve medication adherence. J Adv Nurs. 2014 Sep;70(9):1932-1953. doi: 10.1111/jan.12400. Epub 2014 Apr 1. PMID 24689978
- [Background] Nyandindi U, Palin-Palokas T, Milen A, Robison V, Kombe N, Mwakasagule S. Participation, willingness and abilities of school-teachers in oral health education in Tanzania. Community Dent Health. 1994 Jun;11(2):101-4. PMID 8044706
- [Background] de Silva-Sanigorski A, Ashbolt R, Green J, Calache H, Keith B, Riggs E, Waters E. Parental self-efficacy and oral health-related knowledge are associated with parent and child oral health behaviors and self-reported oral health status. Community Dent Oral Epidemiol. 2013 Aug;41(4):345-52. doi: 10.1111/cdoe.12019. Epub 2012 Nov 17. PMID 23157162
- [Background] Sharma R, Hebbal M, Ankola AV, Murugabupathy V. Mobile-phone text messaging (SMS) for providing oral health education to mothers of preschool children in Belgaum City. J Telemed Telecare. 2011;17(8):432-6. doi: 10.1258/jtt.2011.110416. Epub 2011 Oct 24. PMID 22025742
- [Background] Hall AK, Cole-Lewis H, Bernhardt JM. Mobile text messaging for health: a systematic review of reviews. Annu Rev Public Health. 2015 Mar 18;36:393-415. doi: 10.1146/annurev-publhealth-031914-122855. PMID 25785892
- [Background] Castilho AR, Mialhe FL, Barbosa Tde S, Puppin-Rontani RM. Influence of family environment on children's oral health: a systematic review. J Pediatr (Rio J). 2013 Mar-Apr;89(2):116-23. doi: 10.1016/j.jped.2013.03.014. PMID 23642420
- [Background] Folayan MO, Kolawole KA, Oyedele T, Chukwumah NM, Onyejaka N, Agbaje H, Oziegbe EO, Oshomoji OV. Association between knowledge of caries preventive practices, preventive oral health habits of parents and children and caries experience in children resident in sub-urban Nigeria. BMC Oral Health. 2014 Dec 16;14:156. doi: 10.1186/1472-6831-14-156. PMID 25516332